CLINICAL TRIAL: NCT03592875
Title: Protocol for the Evaluation of Knowledge and Practices in the Systematization of Nursing Care: a Qualitative Research
Brief Title: Evaluation of Knowledge and Practices in the Systematization of Nursing Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Luiz Carlos de Abreu (Other)
Responsible Party: Sponsor-Investigator, Luiz Carlos de Abreu, Assiciated Professor, Faculdade de Medicina do ABC
Organization: Faculdade de Medicina do ABC (Other)
Other Study IDs: 48259915.1.0000.5009
Record Dates: First submitted 2018-07-10; First posted 2018-07-19 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Nursing Personnel
MeSH Terms: interventions — Nurses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Professional nurses: A semi-structured interview will be used for data collection with 16 guiding questions addressing aspects related to Nursing Care Systematization knowledge and practices.
  Interventions: Behavioral: Professional nurses

INTERVENTIONS:
Behavioral: Professional nurses — The nurses will be interviewed by a semi-structured guiding with 16 questions addressing aspects related to Nursing Care Systematization knowledge and practices.

SUMMARY:
Objective to analyse the performance of nurses in the implementation of Nursing Care Systematization - (NCS). This Study is a descriptive research developed from a qualitative approach. The content analysis must be developed through three chronological poles allowing the researcher to construct an analysis structure that corresponds to the needs of the research and the objectives of the proposed research; The chronological poles of content analysis are described as: Phase 1 - Pre-analysis, Phase 2 - Exploration of the material: Phase 3 - Treatment of the results obtained and interpretation. Only a semi-structured interview will be conducted with the research subjects who meet the inclusion criteria of the study, preserving the identity of the individuals and guaranteeing the right to quit the research at any time during the interview.

DETAILED DESCRIPTION:
Study design

It is a descriptive research developed from a qualitative approach. The descriptive study will allow to accurately present facts or phenomena of the studied reality.

The qualitative approach, according to Minayo (2010), arises from the impossibility of investigating and understanding by mean of statistical data some phenomena focused on perception, intuition and subjectivity. Through qualitative evaluation will be exposed experience and common sense through the actions of understanding, interpreting and promoting the dialectics necessary for understanding.

Research scenario

The implementation of this research protocol will be performed at Hospital of Rio Branco - HUERB, an institution maintained by the state public administration, linked to the State Health Secretariat, a member of the Unified Health System (SUS). The mission of HUERB is to provide humanized care with quality and ethics, respecting socio-cultural diversity to all who seek an emergency care service.

This emergency service attends clinical emergencies, surgical and traumatic in adults and children, with back up beds in medical clinic, treatment of acute intoxication and alcohol and other drug withdrawal, paediatric emergency, surgical centre and service of intensive care unit. Altogether there are two hundred and four beds distributed between beds of hospitalization, observation and emergency.

This component of the Urgency and Emergency Network is one of the entry points for secondary level of health care and is a reference for the entire State of Acre, Brazil, and border countries, Bolivia and Peru.

Study participants

Will be part of the set of research participants the professional nurses who perform assistance activities in Hospital of Rio Branco- HUERB at the Emergency Hospital of Rio Branco. It is estimated 30 interviews that will be consolidated by the saturation method.

Collection instrument of empirical material

A semi-structured interview will be used for data collection with 16 guiding questions addressing aspects related to NCS knowledge and practices.

The semi-structured interviews will valorise the researcher's presence and offer all possible perspectives to reach the spontaneity necessary for qualitative research. The interviews start from certain questions that are not born a priori, but from information that the researcher already has about the phenomenon that is of interest to study. In this sense, the informant will have the freedom to follow the line of his thought and his experiences within the main focus placed by the investigator.

Process of Saturation, Corpus Organization and Data Analysis

The organization of the chronological poles will be carried out according to the technique of Content Analysis (CA) through stages that will enable to describe and interpret the subjects' speeches (Bardin, 2009).

According to Bardin (2009) the content analysis must be developed through three chronological poles allowing the researcher to construct an analysis structure that corresponds to the needs of the research and the objectives of the proposed research;

* Phase 1 - Pre-analysis: stage of the organization itself. In it the documents that will be submitted for analysis are selected, the hypotheses and the objectives are formulated and the rules that base the final interpretation are elaborated.
* Phase 2 - Material exploration: this stage consists essentially of coding, discount or enumeration operations, according to pre-formulated rules. It constitutes the identification of the units of record, units of context and subjects that arise from the readings. In this stage, the thematic units and registration units of this study will be identified. It is emphasized that the thematic categories that were explored in this phase will be built focused on the objectives in the previous phase.
* Phase 3 - Treatment of results obtained and interpretation: the gross results will be treated in a way that in the end has a meaning. At this stage, the investigator may propose inferences and advance interpretations about the intended objectives or relate to other unexpected discoveries.

For the completion of data collection (conducting interviews) the researcher will consider the process of saturation of the speeches of the subjects which consists in analysing the empirical data that will be collected. The investigator should focus on the perception of the decrease of new information in each interview, considering the saturation point when the new interviews do not present additions or insignificant information to the research directed by the objectives of the protocol.

Following the steps proposed by Bardin in the pre-analysis the researcher will transcribe the interviews that will allow the floating reading necessary for the initial organization of CORPUS (set of documents that will be exposed to the analysis) that will be analysed; Reaffirmed the objectives of the study, that are: understand the nurses' perception about NCS; Describe the panorama of nursing professional performance in a hospital environment without NCS; Identify in nurses' practices elements that are consistent with the NCS; and identify elements that hinder the NCS implementation process.

Based on the objectives of the study, the researcher predetermined the thematic categories named as:

1. Daily practices in assistance;
2. The NCS Knowledge;
3. Difficulties to implement the NCS;
4. The NCS training and
5. The NCS importance. Thus, to determine the end of the collection, the saturation process will be used; the researcher should consider the convergence of the respondents' speeches considering the categories mentioned above.

For the development of the content analysis is oriented the codification of textual fragments called record units (RU) and subsequent construction of the called context units (CU) that provide sensing to the speeches of respondents; for the implementation of the codification, in the material exploration stage, rules were defined for the systematic development of the enumeration and codification of the registration units by the researcher. The default rules were:

Define representative colours for each category: Category 1 = YELLOW; Category 2 = RED; Category 3 = GREEN; Category 4 = BLUE; and category 5 = PINK;

1. Cut the UR by marking the colour of the representative category;
2. Use the weighted frequency method to determine the representativeness of the categories in the subjects' speeches;
3. To evaluate the URs of NCS KNOWLEDGE using the intensity and direction method through the bipolar scale;
4. Construct the CU using as reference the RUs and inferences arising from the exploration of the material.

Figure 1 presents the flowchart of the construction of the pre-analysis and structuring of CORPUS for content analysis.

After all the reasoning of the rules and how the researcher will direct their analysis of content, will proceed the second stage called exploration of the material; to begin the rules implementation the researcher should develop a new reading of CORPUS.

The CORPUS in this research will be structured in an excel worksheet composed by the transcription of the answers of the respondents, tables with the registration of RU, CU and analytical categories according to Bardin technique, analytical categories and evidences identified with the analysis, registration of the weighted frequencies of the RUs by category, evaluation of the direction and intensity of the RUs for the NCS KNOWLEDGE category and a synthesis of saturation/category points that determined the closure of the data collection.

In the implementation of the CORPUS reading, the RU/category will be cut using the coloured rule predetermined in the previous step for all the speeches of the subjects interviewed.

The application of the weighted frequency will allow the correct direction of the analysis of each questioning for the thematic categories and the use of the intensity and direction for the RUs referring to the NCS KNOWLEDGE category to define the intensity of the right and wrong answers by the subjects.

The exploration of the material will enable the codification and enumeration of RUs and the construction of CUs, which is the first significant inference for the analysis of the subjects' speech and interpretations made by the researcher. Table I shows an example of how the RU and CU will be organized by analytical category, which is the product of the exploraion phase of the material.

Figure II represents an example of the flow chart of the implementation of the rules described above and the beginning of the organization of the evidences that will be identified until step 2.

In the third stage, called Treatment of the results obtained and interpretation, a revision of the CU will be implemented, finalizing the construction of it and organizing the main evidences raised in step 2 to proceed a later interpretation of the results obtained with the exploration of the material.

In this stage the construction of the table with the categories and a summary of the evidences that will be submitted to the interpretation of the researcher are going to completed and will support the construction of the final report of the results and final discussion of the research in the light of the NCS literature.

ELIGIBILITY:
Inclusion Criteria:

* nurses who are at the Emergency of Hospital of Rio Branco - HUERB
* agree to participate in the interview and who sign the Informed Consent Form - ICF

Exclusion Criteria:

* none

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: nurses who are at the Emergency of Hospital of Rio Branco - HUERB
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Nurses' knowledge about Nursin Care Systematization | 2 months
  Nurses' knowledge will be evaluated through the semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Italla MP Bezerra, Ph.D., Principal Investigator — EMESCAM

IPD SHARING:
Plan to Share IPD: Undecided